CLINICAL TRIAL: NCT01379911
Title: Developing and Validating a Method for Satiety Studies
Brief Title: Developing Methods for Completing Future Satiety Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amy Tucker, Manager, HNRU, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11AP036
Record Dates: First submitted 2011-06-15; First posted 2011-06-23 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Lack of Satiety
Keywords: Satiety; Food intake; Yogurt
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yogurt with added inulin (Active Comparator): Yogurt with 6g of added inulin
  Interventions: Other: Yogurt
- Regular yogurt (Placebo Comparator): Regular yogurt without added inulin
  Interventions: Other: Yogurt

INTERVENTIONS:
Other: Yogurt

SUMMARY:
Satiety is defined as the inhibition of eating, as a consequence of fullness after consuming food. Being able to effectively measure satiety is an important concept that has implications in the treatment and prevention of overweight and obesity. Increasing post-meal satiety is recognized a useful strategy for weight management. Recently, the category of foods marketed as having satiating effects has seen significant growth and this trend is expected to continue. The purpose of this project is to develop and validate methods for assessing the degree of satiety induced by foods and natural health products using commercially available food products.

This trial will examine the effects of a commercially available yogurt (containing added protein and fibre) on self-reported satiety and hunger, as well as food intake in both controlled and uncontrolled settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women with regular hormonal contraceptive use, aged between 20 and 35 years
* BMI of 20.0-24.9 kg/m2
* Regular yogurt consumers (i.e. > 3 servings per week)

Exclusion Criteria:

* Taking any regular medications or herbal supplements other than a multivitamin or folic acid supplement.
* History of cardiovascular disease (including hypertension), diabetes, hypoglycemia, gum disease or any other medical condition
* Vegans or vegetarians who exclude dairy products
* Milk allergies or any other food allergies
* Anyone with known anaphylactic allergic reactions, food or otherwise
* Dislike or unwillingness to consume study foods
* Gastrointestinal disease or disorders, including Celiac disease, lactose intolerance, irritable bowel syndrome, etc.
* BMI <20.0 or > 25.0 kg/m2
* Current participation in diet/weight-loss programs and/or changes of > 5 kg body weight within the past 6 months
* Unusual dietary patterns (i.e. routinely skipping breakfast or other meals)
* Unusual sleep patterns (i.e. shift workers)
* High habitual intake of caffeinated beverages or alcohol
* Restrained or disinhibited eaters, defined by the Three Factor Eating Questionnaire
* Smokers

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Self-reported ratings of satiety | Outcome measures will be assessed at fasting (0 min) and postprandially (every 30 min) for 3 hours.
  The study consists of two trial days (pre- and post home consumption) per study period, one for each of 2 yogurts. Each study visit involves a 4-hour stay at the HNRU. The pre-study visit will be followed by a 6-day yogurt self-administration period where participants will consume the assigned yogurt at breakfast. Thus, the acute satiety effects of the yogurts will be replicated in a controlled (laboratory) setting and evaluated over a 6-day period in an uncontrolled (home/lifestyle) environment.

SECONDARY OUTCOMES:
Food intake | One week
  Study will include food and caloric intake over entire study day and for 6 days subsequent to initial study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Wright, Ph.D., Principal Investigator — University of Guelph
Locations (1):
- Human Nutraceutical Research Unit, University of Guelph, Guelph, Ontario, Canada